CLINICAL TRIAL: NCT02725814
Title: Sucrose Practices for Pain in Neonates Part B: Efficacy of Repeated Sucrose Administration, Infant Response to Administration, and Effect on Outcomes
Brief Title: Sucrose Practices for Pain in Neonates Part B
Acronym: SPiN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); IWK Health Centre (Other); The Ottawa Hospital (Other); Children's Hospital of Eastern Ontario (Other)
Responsible Party: Principal Investigator, Bonnie Stevens, Associate Chief of Nursing Research, Senior Scientist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: REB1000051066; 126167 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2016-03-09; First posted 2016-04-01 (Estimated); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Pain
Keywords: Sucrose; Effectiveness; Healthcare Delivery; Neonates; Nursing
MeSH Terms: conditions — Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sucrose (Experimental)
  Interventions: Other: 24% Sucrose Solution

INTERVENTIONS:
Other: 24% Sucrose Solution — Two minutes prior to the start of a painful procedure neonates will receive 0.12ml of 24% sucrose solution, over a period of no more than 1 minute. A pacifier will be offered immediately following sucrose administration for non-nutritive sucking if the infant is able to hold the pacifier securely. The sucrose study dose is to be repeated as needed based on pain response and procedure duration.

SUMMARY:
Recent studies show that babies in hospital undergo an average of 4 to 5 painful procedures, such as heel lances, every day. Sucrose (sugar water) has been shown to be effective for reducing babies' pain during painful procedures. Unfortunately, sucrose is not used as often as it could be to reduce babies' pain. This may be due to lack of certainty about the least effective amount of sucrose to use and concerns about the long-term effects of repeated use of sucrose on infant development. Factors within the hospital units where babies receive care may also influence caregivers' decisions to use sucrose. In this research the investigators will conduct two main studies. In the first study the investigators determined the lowest amount of sucrose needed to manage babies' pain effectively. In the second study the investigators will explore (a) if this amount of sucrose can manage pain when it is used repeatedly for all painful procedures while the baby is hospitalized and (b) whether consistent use of sucrose influences the development of babies when they are 18 and 36 months old. During the second study, the investigators will also examine the hospital units where the babies receive care. They will look at staff support for research, time and resources and other factors that promote and prevent sucrose use. The results of these studies will be used to determine the best management of babies' pain during painful procedures in hospitals to achieve the best outcomes.

ELIGIBILITY:
Inclusion:

* less than 32 weeks gestational age at birth
* admitted to the neonatal intensive care unit (NICU)
* expected to have heel lances for routine blood tests
* yet to reach 10 days of life at the time of study enrollment.

Exclusion:

* known hypersensitivity to sucrose, corn, corn products or any component of the formulation
* short-bowel syndrome
* carbohydrate intolerance
* unable to swallow/absent gag reflex (e.g., pharmacologically muscle relaxed, unconscious, or heavily sedated)

Max Age: 10 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 172 (Actual)
Dates: Start 2016-03; Primary Completion 2022-04 (Actual); Study Completion 2022-04 (Actual)

PRIMARY OUTCOMES:
Pain intensity | Measured 30 seconds post-painful procedure. (NB: Enrolled infants may be evaluated for multiple painful procedures.)
  Assessed by the Premature Infant Pain Profile - Revised (PIPP-R)
Pain intensity | Measured 60 seconds post-painful procedure. (NB: Enrolled infants may be evaluated for multiple painful procedures.)
  Assessed by the Premature Infant Pain Profile - Revised (PIPP-R)
Neurodevelopment (cognitive, language and motor development) | 18 months corrected gestational age
  Assessed by the Bayley Scales of Infant and Toddler Development (BSITD-III)
Neurodevelopment (cognitive, language and motor development) | 36 months corrected gestational age
  Assessed by the Bayley Scales of Infant and Toddler Development (BSITD-III)
Neurodevelopment (social-emotional functioning) | 36 months corrected gestational age
  Assessed by the Ages & Stages Questionnaires: Social-Emotional, Second Edition (ASQ:SE-2)
Neurodevelopment (vision, hearing, speech, emotion, dexterity, self-care, cognition, pain, general health and behaviour) | 36 months corrected gestational age
  Assessed by the Health Status Classification System-Preschool (HSCS-PS)

CONTACTS AND LOCATIONS:
Overall Officials: Bonnie Stevens, PhD, Principal Investigator — The Hospital for Sick Children
Locations (5):
- Canada (5):
  - IWK Health Centre, Halifax, Nova Scotia
  - Children's Hospital of Eastern Ontario, Ottawa, Ontario
  - The Ottawa Hospital, Ottawa, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - The Hospital for Sick Children, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bueno M, Ballantyne M, Campbell-Yeo M, Estabrooks C, Gibbins S, Harrison D, McNair C, Riahi S, Squires J, Synnes AR, Taddio A, Victor C, Yamada J, Stevens B. Cumulative sucrose exposure for repeated procedural pain in preterm neonates and neurodevelopment at 18 months of corrected age: a prospective observational longitudinal study. BMJ Paediatr Open. 2024 Jul 10;8(1):e002604. doi: 10.1136/bmjpo-2024-002604. PMID 38986541